CLINICAL TRIAL: NCT01622439
Title: Valproate as First Line Therapy in Combination With Rituximab and CHOP in Diffuse Large B-cell Lymphoma
Acronym: VALFRID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Valcuria (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version1.1
Record Dates: First submitted 2012-06-12; First posted 2012-06-19 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2016-09

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Lymphoma; Diffuse large B-cell lymphoma; Valproate; R-CHOP; CD 20
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Valproic Acid; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single, open labeld. (Experimental)
  Interventions: Drug: Valproate; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Valproate — Valproate is given in escalating doses to establish maximum tolerable dose when given together with standard treatment in patients with diffuse large B-cell lymphoma; this is the phase I part of the study. When maximum tolerable dose is established, this dose will be given to remaining patients in the phase II part of the study.
Drug: Rituximab — Vill be given intravenously, 375 mg/m2, every second or third week depending on cycle length (14 or 21 days), for a total of 6 cycles.
Drug: Cyclophosphamide — Vill be given intravenously, 750 mg/m2, every second or third week depending on cycle length (14 or 21 days) for a total of 6 cycles.
Drug: Doxorubicin — Vill be given intravenously, 50 mg/m2, every second or third week depending on cycle length (14 or 21 days), for a total of 6 cycles.
Drug: Vincristine — Vill be given intravenously, 1.2 mg/m2, every second or third week depending on cycle length (14 or 21 days), for a total of 6 cycles.
Drug: Prednisone — Vill be given orally, 50 mg/m2, day 1-5 every cycle, for a total of 6 cycles.

SUMMARY:
Patients with previously untreated diffuse large B-cell lymphoma will receive standard treatment with R-CHOP (rituximab,cyclosphosphamide, doxorubicin, vincristine, and prednison) for 6 cycles, cycle length is 14 or 21 days. In addition, valproate is given three times daily day 1-3 in escalated doses. The rationale for adding valproate to standard treatment is invitro data indicating a sensitizing effect to chemotherapy, and an increase in CD 20-expression.

Patients are included in 3+3 cohorts with escalation of valproate dose, planned dos levels are 30, 60, 80, 100, 120, 140 mg/kg/day. A total of 20 patients will be treated at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Histologically confirmed (according to the WHO classification) diffuse large B-cell lymphoma stage II-IV
* No previous treatment for lymphoma. Corticosteroids for alleviation of lymphoma associated symptoms are allowed
* WHO performance status 0-2
* HIV negativity
* Seronegativity for HCV, HBsAg, anti-HBc, or other active infection uncontrolled by treatment
* Absence of psychiatric illness or condition which could interfere with the subjects ability understand the requirements of the study
* Absence of neurological or neuropsychiatric disorder, interfering with the requirements of the study
* Absence of hearing impairment > grade 2
* Absence of porphyria
* In females: absence of pregnancy and lactation
* All subjects must agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy
* All subjects must agree not to share study medication with another person, and to return all unused study drug to investigators
* Written informed concent according to ICH/GCP and Swedish regulations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Establishment of maximum tolerable dose of valproate. | Participating patients will be followed during study treatment (6 cycles of chemotherapy); 12 weeks or 18 weeks depending on cycle length (14 or 21 days).

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jerkeman, MD, PhD, Principal Investigator — Skåne University Hospital, Dept. of Oncology
Locations (1):
- Skåne University Hospital, Dept. of Oncology, Lund, Sweden

REFERENCES:
- [Derived] Drott K, Hagberg H, Papworth K, Relander T, Jerkeman M. Valproate in combination with rituximab and CHOP as first-line therapy in diffuse large B-cell lymphoma (VALFRID). Blood Adv. 2018 Jun 26;2(12):1386-1392. doi: 10.1182/bloodadvances.2018019240. PMID 29903707